CLINICAL TRIAL: NCT03630042
Title: A Phase II Trial to Investigate the Safety and Efficacy of Rituximab and Pembrolizumab in Relapsed/Refractory Waldenström's Macroglobulinaemia
Brief Title: Investigating the Safety and Efficacy of Rituximab and Pembrolizumab in Relapsed/Refractory Waldenström's Macroglobulinaemia
Acronym: PembroWM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/18/0131; 2018-001767-23 (EudraCT Number); MISP # 56775 (Other Grant/Funding Number: Merck, Sharp & Dohme Ltd)
Record Dates: First submitted 2018-07-13; First posted 2018-08-14 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Waldenstrom Macroglobulinemia
Keywords: Waldenstrom Macroglobulinemia; Relapsed; Refractory; Rituximab; Pembrolizumab
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Recurrence | interventions — pembrolizumab; Rituximab

STUDY DESIGN:
Intervention Model Description: A single arm, non randomised phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab and Rituximab (Experimental)
  Interventions: Drug: Pembrolizumab; Drug: Rituximab

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg IV dose given on day 1 of a three week cycle
Drug: Rituximab — 375 mg/m2 IV dose given up to 8 times in the trial

SUMMARY:
This study is for patients who have previously been treated for Waldenström's macroglobulinaemia (WM) and their disease has either not responded (known as refractory disease) or has returned (known as relapsed disease). Through this study, the researchers would like to find out whether treating these patients with drugs called rituximab and pembrolizumab is a safe and effective combination for this disease.

In this study, pembrolizumab and rituximab will be given together. In other studies pembrolizumab has been shown to be effective at treating diseases similar to WM. The researchers want to test whether giving pembrolizumab and rituximab together is safe and effective.

ELIGIBILITY:
Inclusion criteria

1. Patients ≥18 years old
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
3. Presence of measurable disease, (defined as a serum IgM level of >0.5g/L) and fulfils other World Health Organisation (WHO) diagnostic criteria for WM
4. Relapsed or refractory WM who have received ≥1 prior lines of therapy
5. Adequate renal function: estimated creatinine clearance ≥ 30ml/min as calculated using the Cockroft-Gault equation
6. Adequate liver function, including:

   * Bilirubin ≤1.5x the upper limit of normal (ULN)
   * Aspartate or alanine transferase (AST or ALT) ≤2.5 x ULN
7. Adequate organ and bone marrow function:

   * Neutrophils ≥0.75x109/L
   * Platelets ≥50x109/L
8. Willing to comply with the contraceptive requirements of the trial
9. Negative serum or highly sensitive urine pregnancy test for women of childbearing potential (WOCBP)
10. Written informed consent

Exclusion criteria

1. Refractory to rituximab as defined by progression on/within 6 months of finishing a rituximab based regimen
2. Women who are pregnant or breastfeeding, or males expecting to conceive or father children at any point from the start of treatment until 4 months after the last administration of pembrolizumab
3. Clinically significant cardiac disease within 6 months prior to registration including unstable angina or myocardial infarction, uncontrolled congestive heart failure (NYHA class III-IV), and unstable arrhythmias requiring therapy, with the exception of extra systoles or minor conduction abnormalities. Stable and controlled atrial fibrillation is not an exclusion.
4. History of significant cerebrovascular disease in last 6 months
5. Known central nervous system involvement of WM
6. Clinically significant active infection requiring antibiotic or antiretroviral therapy (including Hepatitis B, C or human immunodeficiency virus (HIV))
7. Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
9. Active autoimmune disease apart from:

   * Type I diabetes or thyroid disease, controlled on medication
   * Skin conditions such as psoriasis, vitiligo or alopecia not requiring systemic treatment
   * Auto-immune thrombocytopenia, thought to be secondary to WM, provided that platelet count meet the criteria specified above, on daily doses of corticosteroid ≤10mg prednisolone or equivalent
10. Prior history of haemolytic anaemia (either warm or cold)
11. History of colitis
12. History of (non-infectious) pneumonitis that required steroids or has current pneumonitis
13. Systemic anti-cancer therapy within 4 weeks prior to trial registration (except for BTK inhibitors, which may continue until cycle 1, day 1 of trial treatment)
14. Received a T cell depleting antibody (e.g. Campath) within 3 months prior to starting treatment
15. Received a live vaccine within 30 days prior to starting treatment
16. Chronic or ongoing active infectious disease requiring systemic treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active hepatitis
17. Patients who have received treatment with any non-marketed drug substance or experimental therapy within 4 weeks prior to starting treatment (unless prior agreed with the TMG)
18. Patients known or suspected of not being able to comply with a study protocol (e.g. due to alcoholism, drug dependency or psychological disorder)
19. Positive serology for Hepatitis B defined as a positive test for HepB surface antigen (HBsAg). Note: patients who are HepB core antibody (HBcAb) positive will only be eligible for the study if the HepB virus deoxyribonucleic acid (HBV DNA) test is negative and patients are willing to undergo monthly monitoring for HBV reactivation
20. Major surgery within 4 weeks prior to trial registration
21. Prior therapy with an anti-PD-1,anti-PD-L1 or CTLA4 monoclonal antibody
22. Prior allogeneic bone marrow transplantation
23. Diagnosis of prior immunodeficiency or organ-transplant requiring immunosuppressive therapy or known HIV or acquired immunodeficiency syndrome (AIDS)-related illness
24. Current or prior use of immunosuppressive therapy within 7 days prior to start of treatment except the following: intranasal, inhaled, topical steroids or local steroid injections (eg. Intra-articular injections); systemic corticosteroids at physiologic doses (<10mg/ day of prednisolone or equivalent)
25. Known or suspected hypersensitivity to components of pembrolizumab and/or rituximab (or other CD20 monoclonal antibody)
26. Current participation in any other clinical trial of an investigational medicinal product (CTIMP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2024-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaimal Kothari, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (9):
- United Kingdom (9):
  - Derriford Hospital, Univeristy Hospitals Plymouth NHS Trust, Plymouth, Devon
  - Torbay and South Devon NHS Foundation Trust, Torquay, Devon
  - Royal Bournemouth Hospital, University Hospitals Dorset NHS Foundation Trust, Bournemouth, Dorset
  - St Bartholomew's Hospital, Barts Health NHS Trust, London, Greater London
  - UCLH, Univeristy College London Hospitals NHS Foundation Trust, London, Greater London
  - The Christie Hospital, The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - Churchill Hospital, Oxford Univeristy NHS Foundation Trust, Oxford, Oxfordshire
  - Bristol Haematology & Oncology Medical Centre, University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - Norfolk and Norwich University Hospital, Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab and Rituximab
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab and Rituximab
Number analyzed (Participants) | 17
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70.4 [64.5 to 76.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status
  0: Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair
  5. Dead
  Participants
    ECOG 0 | 9
    ECOG 1 | 7
    ECOG 2 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving at Least a Major Response Rate at 24 Weeks Post Commencing Treatment
Description: The primary outcome is the percentage of patients achieving at least a major response rate at 24 weeks post commencing treatment. A major response rate is defined as a greater than 50% reduction in paraprotein measurement - this is in line with international recognised response criteria for the disease under investigation. In this single arm study all patients receiving treatment were considered applicable for endpoint analysis. There is no comparison as there is only one arm.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab and Rituximab
Number analyzed (Participants) | 17
Participants | 8

2. Secondary Outcome: Safety and Tolerability of Pembrolizumab and Rituximab as Assessed by the Frequency of Serious and Non-serious Adverse Events, According to CTCAE v5.0
Description: As assessed by the number and grade of serious and non-serious adverse events, graded according to CTCAE v5.0
Time Frame: until 5 months post last IMP administration
Reporting Status: Not Posted

3. Secondary Outcome: Complete Response Rate at 24 Weeks Post Commencing Treatment
Time Frame: 24 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Very Good Partial Response Rate at 24 Weeks Post Commencing Treatment
Time Frame: 24 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Time to Maximal Response as Determined by the Time of Registration to the Maximal Disease Response
Time Frame: Assessed at 12 weeks, 24 weeks and 1 year after commencing treatment
Reporting Status: Not Posted

6. Secondary Outcome: Time to Next Treatment
Description: as determined by the time from registration to the next line of therapy
Time Frame: Assessed once per year after completing treatment (average of 1 year)
Reporting Status: Not Posted

7. Secondary Outcome: Progression Free Survival (PFS) at 1 and 2 Years
Time Frame: 1 and 2 years post commencing treatment
Reporting Status: Not Posted

8. Secondary Outcome: Overall Survival (OS) at 1 and 2 Years
Time Frame: 1 and 2 years post commencing treatment
Reporting Status: Not Posted

9. Secondary Outcome: Quality of Life - Change in Quality of Life (QoL) at 24 Weeks Post Commencing Treatment as Assessed by EORTC QLQ-C30 Questionnaire
Description: Change in quality of life (QoL) at 24 weeks post commencing treatment as assessed by EORTC QLQ-C30 questionnaire. Daily activities and thoughts/feelings experienced by the patient over the week preceding questionnaire completion are graded on a scale from '1-not at all' to '4-very much'. Also rating of overall health and quality of life from '1-very poor' to '7-excellent'
Time Frame: 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Between informed consent and 5 months post last IMP administration.
Arm/Group | Pembrolizumab and Rituximab
All-Cause Mortality (participants affected / at risk) | 5/17
Serious Adverse Events (participants affected / at risk) | 10/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab and Rituximab (N=17)
Fatigue (General disorders) | 1
Fever (General disorders) | 3
Covid-19 (Infections and infestations) | 2
Infection (unknown origin) (Infections and infestations) | 2
Lung infection (Reproductive system and breast disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2
Vaccination complication (Injury, poisoning and procedural complications) | 1
Creatinine increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Stroke (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab and Rituximab (N=17)
Neutropenia (Blood and lymphatic system disorders) | 2
Anemia (Blood and lymphatic system disorders) | 8
Folate deficiency (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Atrioventricular block first degree (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 2
Heart failure with preserved ejection fraction (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Loose stools (Gastrointestinal disorders) | 1
Mouth ulcer (Gastrointestinal disorders) | 1
Chills (General disorders) | 2
Localized edema (General disorders) | 2
Fever (General disorders) | 6
Facial pain (General disorders) | 1
Fatigue (General disorders) | 5
Shoulder pain (General disorders) | 1
Intermittent pain in fingers (General disorders) | 1
Lymph gland infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Thrush (Infections and infestations) | 1
Infection (Infections and infestations) | 2
covid-19 (Infections and infestations) | 2
chest infection (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 7
Platelet count decreased (Investigations) | 2
Weight loss (Investigations) | 1
Creatinine increased (Investigations) | 5
White blood cell decreased (Investigations) | 4
Blood bicarbonate decreased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 4
Serum amylase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 4
Thyroid stimulating hormone increased (Investigations) | 2
White blood cell increased (Investigations) | 2
Platelet count increased (Investigations) | 1
Increased neutrophils (Investigations) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 3
Iron deficiency (Metabolism and nutrition disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Polymylagia rheumatica (Musculoskeletal and connective tissue disorders) | 1
Excision of basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma trunk (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 3
Paresthesia (Nervous system disorders) | 2
Stroke (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Peripheral neuropathy (Nervous system disorders) | 2
Sciatica pain (right leg) (Nervous system disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Other/hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 4
Flushing (Vascular disorders) | 1
Skin lesion (forehead) (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The sample size of 42 was not reached so limited conclusions can be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT03630042/Prot_SAP_000.pdf